CLINICAL TRIAL: NCT00865007
Title: A Phase IV-III Comparative, Randomized, Open-label Study to Evaluate the Efficacy for the Recovery of Peripheral Fat (or of the Extremities) of Lopinavir/Ritonavir in Monotherapy Versus Abacavir/Lamivudine and Lopinavir/Ritonavir
Brief Title: Lopinavir/r Monotherapy Versus Abacavir/Lamivudine and Lopinavir/r for Limb Fat Recovery in Persons With Lipoatrophy
Acronym: KRETA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion SEIMC-GESIDA (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GESIDA-6008; 2008-003748-12 (EudraCT Number)
Record Dates: First submitted 2009-03-18; First posted 2009-03-19 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: HIV Infection; Lipodystrophy; HIV Infections
Keywords: Lipodystrophy; treatment experienced
MeSH Terms: conditions — HIV Infections; Lipodystrophy | interventions — Lopinavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Monotherapy group (Experimental): Lopinavir/ritonavir (LPV/r).
  Interventions: Drug: Monotherapy (Lopinavir/ritonavir)
- Triple arm (Active Comparator): Lopinavir/ritonavir (LPV/r)+ ABC/3TC
  Interventions: Drug: Monotherapy (Lopinavir/ritonavir); Drug: Monotherapy (Lopinavir/ritonavir) + ABC/3TC

INTERVENTIONS:
Drug: Monotherapy (Lopinavir/ritonavir) — NRTI sparing
Drug: Monotherapy (Lopinavir/ritonavir) + ABC/3TC — NRTI sparing regimen
  Arms: Triple arm

SUMMARY:
The aim of this study is to evaluate the efficacy for the recovery of peripheral fat of lopinavir/ritonavir in monotherapy versus abacavir/lamivudine and lopinavir/ritonavir in subjects who developed lipoatrophy while receiving zidovudine plus lamivudine plus abacavir.

DETAILED DESCRIPTION:
After more than ten years since it was started, it has already been established that highly-active antiretroviral treatment (HAART) has caused a dramatic reduction in the morbidity and mortality of human immunodeficiency virus (HIV) infection. However, HAART is not exempt of limitations, namely, its toxicity in the long-term; this is of special importance now that treatment of HIV is chronic.

Most common HAART involves the use of two nucleoside reverse transcriptase inhibitors (nucleoside or nucleotide analogues, NRTIs) and either a protease inhibitor (PI) or a non-analogue reverse transcriptase inhibitor (NNRTI). However, there are other regimens that remove some of these families, such as those based on three NRTIs, ZDV+3TC+ABC.

HAART has been associated with a constellation of major metabolic adverse events, such as fat redistribution (lipodystrophy, lipoatrophy, lipohypertrophy-central obesity - or both) and hyperlipidemia (hypercholesterolemia and hypertriglyceridemia).

Lipoatrophy, specifically, occurs as a loss of subcutaneous fat mass in the upper and lower extremities, with the possible appearance of venomegaly in face and buttocks Lipoatrophy is particularly distressing not only for itself, but for its stigma component, affecting the quality of life and the psychological condition of the patient.This also has a direct impact on treatment compliance, that is reduced, and, therefore, at risk that the therapeutic regimen fails to be effective for resistances selection.

Although initially most metabolic adverse events were attributed to PIs, in recent years it has been shown that lipoatrophy specifically is related more to therapy with NRTIs than with PIs; specifically, d4T, ddI and ZDV.

One of the accepted strategies for the management of lipoatrophy in patients receiving therapy with ZDV is its replacement by other NRTI such as TDF or ABC, and consequently, a significant fat recovery is seen.

In a study where therapy with ZDV was discontinued and continued with NNRTIs (lopinavir/ritonavir-LPV/r and nevirapine-NVP) therapy, fat recovery in the extremities seemed to be higher than in patients where ZDV was replaced by ABC.

Lopinavir (ABT-378) is a potent protease inhibitor of HIV. The proven efficacy and safety of LPV/r-based HAART has led to its inclusion since 2003 in therapeutic guidelines as therapy of preferential start PI/r based.

With regard to its relationship with lipoatrophy, recent data have shown that LPV/r has a low risk induction profile.

In recent years data have been published on the use of LPV/r monotherapy: starting, and induction-maintenance after therapy with HAART with sustained undetectability for at least 6 months.

Given the aforementioned data, in those patients developing lipoatrophy while treated with ZDV+ABC+3TC, the approach of switching to a regimen in the absence of LPV/r-based nucleosides could be even more beneficial than just removing ZDV and maintaining them on a HAART containing LPV/r+ABC+3TC. Despite the fact that lipoatrophy associated with ABC/3TC is very low in treatment-naive patients, it has yet to be demonstrated that discontinuing even "benign" nucleosides could provide an additional benefit in patients that had already developed lipoatrophy.

Accordingly, the working hypothesis for this study would be as follows: the recovery or reversion of lipoatrophy would increase in patients receiving LPV/r in monotherapy vs those switching to a classic LPV/r-based HAART. The absence of any nucleoside would then be beneficial for fat recovery in the extremities.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of the willingness of the patient to participate in this study after being informed on all the aspects of the trial that may influence their decision, signing and dating the written informed consent form approved by the Ethics Committee.
* The patient is 18 years of age or older.
* (Documented) HIV-1 infection.
* Receiving treatment with ZDV+3TC+ABC (in continuous antiretroviral treatment, without discontinuation periods, for the past 6 months).
* There is confirmation that during the 6 months prior to inclusion in the study the viral burdens were below 50 copies/mL.
* A viral burden below 50 copies/mL no more than 30 days before starting the study.
* No previous history of virological failure while on antiretroviral treatment with protease inhibitors (PIs). That is, they have never switched protease inhibitors for suspected or documented virological failure. The changes in protease inhibitor due solely to toxicity, simplification or optimization are acceptable.
* Clinical evidence of moderate to severe lipoatrophy (according to the case definition as scoring >- 2. For inclusion in the study, the subject should have moderate to severe lipoatrophy in at least one site, and defined by the physician.
* Absence of signs of acute disease.
* Patient has not been treated for an active opportunistic infection within the 30 days prior to the baseline visit.
* Patient with Karnofsky index >- 70.
* During the study, the patient does not require and agrees not to take any of the following drugs that are contraindicated with LPV/r: astemizole, terfenadine, midazolam, triazolam, cisapride, certain ergot derivatives (ergotamine, dihydroergotamine, ergonovine, methylergonovine), pimozide, propafenone, and flecainide. Rifampin, a potent enzyme inducer, should not be administered with the study medication due to the possibility of a significant decrease in LPV/r concentrations during concomitant administration, nor drugs contraindicated with 3TC and ABC that in principle should not be being taken, as they are part of the treatment at the screening.
* Patient agrees not to take any medication, including over-the-counter medicines, alcohol, drugs, or herbal preparations without the knowledge and approval of the principal investigator.
* Laboratory tests have been performed on the patients in the past 30 days:
* G/dL hemoglobin >8.0
* Absolute neutrophil count 750 cells/microl
* Platelet count 20,000/microl
* ALT or AST <5 x upper normal limit (UNL)
* Creatinine <1. 5 x UNL
* Triglycerides <750 mg/dL.
* For women, a negative result of a pregnancy test is available and they agree to use throughout the study a barrier contraceptive method of proven reliability in the investigator's opinion.

Exclusion Criteria:

* Patients with a history of virological failure on treatment with PIs; that is, that they have at some point switched to PIs for confirmed or documented virological failure.
* Patients with positive serum hepatitis B surface antigen.
* Patients requiring treatment with drugs where combination with LPV/r is contraindicated.
* Presence of active opportunistic disease or wasting syndrome or under antitumoral treatment with chemotherapy.
* Patients treated in the previous 16 weeks with agents susceptible to insulin (glitazones or metformin), anabolic steroids, growth hormone or any agent that could interfere with the study drugs.
* Active drug addiction or psychiatric disease that may prevent protocol compliance. Use of cannabis or being on methadone treatment are excepted, provided protocol compliance is not compromised in the investigator's opinion.
* Pregnant women or nursing mothers, and women of childbearing age if they do not agree to use a barrier contraceptive method throughout the study of proven reliability in the investigator's opinion.
* In the opinion of the principal investigator, the patient is unlikely to comply with the study protocol, or the patient is not eligible for any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2008-12; Primary Completion 2012-06 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Absolute change in limb fat measured by DEXA at 48w | 48 weeks

SECONDARY OUTCOMES:
Absolute change in limb-fat measured by DEXA at 96 weeks | 96 weeks
Lipid changes at Week 24, 48, 72 and 96 | 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jose Ignacio Bernardino, Study Chair — Hospital La Paz; Jose Ramon Arribas, Study Chair — Hospital La Paz
Locations (10):
- Spain (10):
  - Hospital General Universitario de Alicante, Alicante, Alicante
  - Hospital Sant Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Clinico y Provincial, Barcelona, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba, Cordoba
  - Hospital Severo Ochoa, Leganés, Madrid
  - Hospital La Paz, Madrid, Madrid
  - Hospital Doce de Octubre, Madrid, Madrid
  - Hospital Xeral Cies, Vigo, Pontevedra
  - Hospital de Donostia, Donostia / San Sebastian, San Sebastian
  - Hospital de Basurto, Bilbao, Vizcaya

REFERENCES:
- [Derived] Bernardino JI, Pulido F, Martinez E, Arrizabalaga J, Domingo P, Portilla J, Ocampo A, Munoz J, Torres R, Arribas JR; GESIDA-6008-KRETA Study Group. Switching to lopinavir/ritonavir with or without abacavir/lamivudine in lipoatrophic patients treated with zidovudine/abacavir/lamivudine. J Antimicrob Chemother. 2013 Jun;68(6):1373-81. doi: 10.1093/jac/dks540. Epub 2013 Feb 5. PMID 23386261